CLINICAL TRIAL: NCT02742909
Title: Acute Effect of Recombinant Human Brain Natriuretic Peptide in Patients With Pulmonary Hypertension Associated With Acute Exacerbation of Chronic Pulmonary Disease
Brief Title: Acute Effects of rhBNP in Patients With PH Associated With Acute Exacerbation of Chronic Pulmonary Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: LI ZHAO (Other)
Responsible Party: Sponsor-Investigator, LI ZHAO, professor /director, Shengjing Hospital
Organization: Shengjing Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SJHX-001
Record Dates: First submitted 2015-10-09; First posted 2016-04-19 (Estimated); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rhBNP (Active Comparator): the study is a self controlled study. Each patient was studied on two occasions (6 hours apart). One occasion the subject received rhBNP 1.5ug/kg IV bolus followed by an infusion of 0.0075ug/kg/min for 24 hours; other occasion the subject received IV placebo bolus followed by a placebo infusion for 24 hours .these were administered in random order in double blind fashion.The date of this arm is from the occasion the subject received rhBNP.
  Interventions: Drug: rhBNP
- Placebo (Placebo Comparator): the study is a self controlled study. Each patient was studied on two occasions (6 hours apart). One occasion the subject received rhBNP 1.5ug/kg IV bolus followed by an infusion of 0.0075ug/kg/min for 24 hours; other occasion the subject received IV placebo bolus followed by a placebo infusion for 24 hours .these were administered in random order in double blind fashion.The date of this arm is from the occasion the subject received placebo.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: rhBNP — rhBNP was administered as a continuous infusion for 24 hours before or after placebo
  Other Names: Recombinant Human Brain Natriuretic Peptide
  Arms: rhBNP
Drug: placebo — normal saline as a placebo was administered as a continuous infusion for 24 hours
  Other Names: normal saline
  Arms: Placebo

SUMMARY:
To evaluate the acute effect of recombinant human brain natriuretic peptide(rhBNP) on pulmonary hypertension of acute exacerbations of chronic pulmonary disease. rhBNP was administered as a continuous infusion for 24 hours , pulmonary artery pressure and other hemodynamic parameters were monitored by Swan- Ganz catheter.

DETAILED DESCRIPTION:
Pulmonary hypertension (PH) is a descriptive name for abnormally elevated pressures in the pulmonary vasculature, which seriously affects the quality of life and survival of patients. Currently, no effective drugs treatment was used in patients with pulmonary hypertension due to acute exacerbation of lung disease. Recombinant Human Brain Natriuretic Peptide (rhBNP)was approved in 2001 for use in patients with acute heart failure on the basis of studies showing a reduction in pulmonary-capillary wedge pressure(PCWP) and pulmonary arterial pressure (PAP) and improvement cardiac output (CO) . Thus, the study was designed to administer rhBNP as a continuous infusion for 24 hours on pulmonary hypertension of acute exacerbations of chronic pulmonary disease monitoring by Swan- Ganz catheter. Each patient was studied on two occasions (6 hours apart). One occasion the subject received rhBNP 1.5ug/kg IV bolus followed by an infusion of 0.0075ug/kg/min for 24 hours; other occasion the subject received IV placebo bolus followed by a placebo infusion for 24 hours .these were administered in random order in double blind fashion.

ELIGIBILITY:
Inclusion Criteria:

1. age>18 years old, male or female;
2. in acute exacerbation period and with a history of chronic respiratory diseases;
3. cardiac ultrasound showed a pulmonary hypertension ≥50mmHg;
4. grade II or WHO grade of heart function;
5. signed informed consent.

Exclusion Criteria:

1. pulmonary hypertension not associated with chronic lung disease;
2. Acute or severe chronic left heart failure;
3. severe respiratory failure during receipt of non-invasive or invasive ventilator therapy;
4. mPAP≤25mmHg or pulmonary capillary wedge pressure (PCWP) ≥15mmHg at rest as assessed by Swan- Ganz catheter;
5. a high risk of hypotension (systolic pressure <100 mmHg or 110 mmHg with the use of intravenous nitroglycerin);
6. Uncontrolled arterial hypertension;
7. acute coronary syndrome;
8. Severe left ventricular hypertrophy;
9. Congenital or acquired valvular or myocardial disease;
10. end-stage renal disease during receipt of renal replacement therapy;
11. clinically significant anemia;
12. other contraindications for vasodilators;
13. treatment with dobutamine (at a dose ≥5 μg per kilogram of body weight per minute);
14. treatment with milrinone or levosimendan within the previous 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-12; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
pulmonary artery systolic pressure (PASP) measured by Swan-Ganz catheter | baseline , 0.5 hour, 1hour, 2hours, 4hours, 8hours, 12hours, 20hours, 24hours, 27hours and 30hours
  we are going to record a change
pulmonary artery diastolic pressure(PADP) measured by Swan-Ganz catheter | baseline , 0.5 hour, 1hour, 2hours, 4hours, 8hours, 12hours, 20hours, 24hours, 27hours and 30hours
  we are going to record a change
mean pulmonary artery pressure(mPAP) measured by Swan-Ganz catheter | baseline , 0.5 hour, 1hour, 2hours, 4hours, 8hours, 12hours, 20hours, 24hours, 27hours and 30hours
  we are going to record a change
pulmonary vascular resistance(PVR) measured by Swan-Ganz catheter | baseline , 0.5 hour, 1hour, 2hours, 4hours, 8hours, 12hours, 20hours, 24hours, 27hours and 30hours
  we are going to record a change
cardiac output(CO) measured by Swan-Ganz catheter | baseline , 0.5 hour, 1hour, 2hours, 4hours, 8hours, 12hours, 20hours, 24hours, 27hours and 30hours
  we are going to record a change

SECONDARY OUTCOMES:
heat rate (HR) | baseline and 30 hours
respiratory rate(RR) | baseline and 30 hours
blood pressure(BP) | baseline and 30 hours
blood oxygen saturation(SPO2) | baseline and 30 hours
Brog classification | baseline and 30 hours
  this is a classification table for patient' s feeling of fatigue and dyspnea. from 1 to 10 degree.
Brain Natriuretic Peptide(BNP) in blood | baseline and 30 hours
N-terminal pro-Brain Natriuretic Peptide(NT-pro BNP) in blood | baseline and 30 hours
Potential of Hydrogen(PH) in artery blood gas analysis | baseline and 30 hours
arterial partial pressure of oxygen(PaO2) | baseline and 30 hours
arterial partial pressure of carbon dioxide (PaCO2) | baseline and 30 hours
oxygenation index in artery blood gas analysis | baseline and 30 hours
alveolar-arterial oxygen difference in artery blood gas analysis | baseline and 30 hours

CONTACTS AND LOCATIONS:
Overall Officials: LI ZHAO, DOCTOR, Principal Investigator — SHENJING HOSPTIAL OF CHINA MEDICAL UNIVERSITY
Locations (1):
- Shenjing Hospital, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Haeck ML, Vliegen HW. Diagnosis and treatment of pulmonary hypertension. Heart. 2015 Feb;101(4):311-9. doi: 10.1136/heartjnl-2011-301386. Epub 2014 May 22. No abstract available. PMID 24855320
- [Background] O'Connor CM, Starling RC, Hernandez AF, Armstrong PW, Dickstein K, Hasselblad V, Heizer GM, Komajda M, Massie BM, McMurray JJ, Nieminen MS, Reist CJ, Rouleau JL, Swedberg K, Adams KF Jr, Anker SD, Atar D, Battler A, Botero R, Bohidar NR, Butler J, Clausell N, Corbalan R, Costanzo MR, Dahlstrom U, Deckelbaum LI, Diaz R, Dunlap ME, Ezekowitz JA, Feldman D, Felker GM, Fonarow GC, Gennevois D, Gottlieb SS, Hill JA, Hollander JE, Howlett JG, Hudson MP, Kociol RD, Krum H, Laucevicius A, Levy WC, Mendez GF, Metra M, Mittal S, Oh BH, Pereira NL, Ponikowski P, Tang WH, Tanomsup S, Teerlink JR, Triposkiadis F, Troughton RW, Voors AA, Whellan DJ, Zannad F, Califf RM. Effect of nesiritide in patients with acute decompensated heart failure. N Engl J Med. 2011 Jul 7;365(1):32-43. doi: 10.1056/NEJMoa1100171. PMID 21732835
- [Background] Mingguang Huang,Yingjun Dong. Clinical observation on rhBNP in treating patients with pulmonary artery hypertension. Shanxi Medical Journal,2011,40(6):545-546.